CLINICAL TRIAL: NCT01858337
Title: Mum Can I Have Vegetables Again? Development of Vegetable Preferences.
Acronym: VaVo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL28886.081.09
Record Dates: First submitted 2013-05-03; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Vegetable Intake After Weaning With Vegetables or Fruits; Fruit Intake After Weaning With Vegetables or Fruits
Keywords: weaning; infants; vegetables; repeated-exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- green beans group, (Experimental): 1 of the 2 vegetable groups. The infants were weaned only with vegetables. With green beans every other day and another vegetable on the days in between.
  Interventions: Other: green beans group
- Artichoke group (Experimental): 1 of the 2 vegetable groups. The infants were weaned only with vegetables. With Artichoke every other day and another vegetable on the days in between
  Interventions: Other: Artichoke group
- Apple group (Active Comparator): 1 of the 2 fruit groups. The infants were weaned only with fruits. With Apple every other day and other fruits on the days in between
  Interventions: Other: Apple group
- Plums group (Active Comparator): 1 of the 2 fruit groups. The infants were weaned only with vegetables. With Plums every other day and other fruits on the days in between
  Interventions: Other: Plums group

INTERVENTIONS:
Other: green beans group — Infants were weaned with vegetable purees for the first 18 days of weaning. One vegetable type per day. With green beans every other day.
  Arms: green beans group,
Other: Artichoke group — Infants were weaned with vegetable purees for the first 18 days of weaning. One vegetable type per day. With artichoke every other day.
  Arms: Artichoke group
Other: Apple group — Infants were weaned with fruit purees for the first 18 days of weaning. One fruit type per day. With apple every other day.
  Arms: Apple group
Other: Plums group — Infants were weaned with fruit purees for the first 18 days of weaning. One fruit type per day. With Plums every other day.
  Arms: Plums group

SUMMARY:
* Rationale: Despite the health benefits, children's consumption of vegetables is below the recommendations. Most human food preferences are learned through mere exposure, imitation, and conditioning principles. During the last years, it has become clear that the development of food preferences starts very early in life. Furthermore, preferences that are learned early in life, are relatively stable and may track into adulthood. However, it is unclear how vegetable preferences develop from infancy until young childhood. In order to influence vegetable consumption, it is essential to study the opportunities to develop a preference for vegetable products early in childhood.
* Objective: The aim of this study is to investigate the effect of repeated exposure to vegetables compared to repeated exposure to fruit during weaning on short and long term vegetable and fruit intake. Furthermore, the stability of the learned fruit or vegetable preferences and the later food preferences are measured (i.e. vegetable, fruits, sweets).
* Study design:

In this longitudinal study we will measure the development of preferences for a particular vegetable or fruit type within 4 to 6 months old subjects, during a 19 day exposure period to fruit or vegetables (of which 9 days exposure to the target fruit or vegetable) and 6 months after this exposure period. In addition, we compare the food preferences (fruit, vegetable, sweet foods in general), after 6 months, between infants who were weaned with a variety of fruits and infants who were weaned with a variety of vegetables.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 4 and 6 months of age that are apparently healthy are invited to participate in the study. The parents have to give permission for themselves and for their infant to participate by signing an informed consent. By signing the informed consent the parents also agree to participate in the study for 2 years.

Exclusion Criteria:

* The parents will not sign the informed consent
* The parents have already started weaning their child
* The infant has a food allergy or intolerance
* The child has medical problems that influences with eating or food digestion. (e.g. schisis, problems with the bowls)
* The child has a known cognitive or physical developmental problem, which influences how the child's reaction or facial expressions.

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2009-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in Vegetable and fruit intake | At the first 19 days of weaning (4-6 months of age)
  Change in Vegetable and fruit intake from before to after the repeated exposure to it. Measured at day 1 and 2 and day 17 and 18 at the intervention.
Intake of the target Vegetables and fruits at 12 months of age. | 6 months after the intervention. Mean age 12 months.
  Vegetable and fruit intake at 12 months of age. Measured in the lab. Fruit group received apple, plum and green beans at 3 different days
Green beans and Apple intake at 23 months of age. | when infants are 23 months of age
  Green beans and Apple intake at 23 months of age.

SECONDARY OUTCOMES:
Vegetable and in fruit intake after the repeated exposure | After the repeated exposure period during the first 19 days of weaning
  Difference in vegetable intake between vegetable and fruit groups and in fruit intake between the vegetable and fruit groups. Vegetable intake is measured on day 17 and 18 in the vegetable groups and in the fruit groups at day 19 (when fruit groups gets the first vegetable.

CONTACTS AND LOCATIONS:
Overall Officials: Cees de Graaf, Prof., Study Director — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Result] Barends, C.d.V., J; Mojet, J & de Graaf, C, Effects of repeated exposure to either vegetables or fruits on infant's vegetable and fruit acceptance at the beginning of weaning. Food quality and preference, 29 , 157-165, 2013